CLINICAL TRIAL: NCT00307502
Title: Cross-sectional Study for the Characterisation of the Pharmacokinetic Parameters of Protease Inhibitors and Non-nucleoside Analog Reverse Transcriptase Inhibitors in the Spanish Population of HIV-infected Subjects
Brief Title: Study to Determine the Pharmacokinetic Behavior of Antiretroviral Drugs in Patients Infected by HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK-TRANSVERSAL; 2004-001516-32
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: protease inhibitors; non-nucleoside analog reverse transcriptase inhibitors; pharmacokinetic models; treatment experienced; HIV
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; efavirenz; Indinavir; Ritonavir; Nelfinavir; Saquinavir; Lopinavir; lopinavir-ritonavir drug combination; Atazanavir Sulfate; atazanavir, ritonavir drug combination; fosamprenavir; tipranavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- NVP (Experimental): Nevirapine
  Interventions: Drug: Nevirapine
- EFV (Experimental): Efavirenz
  Interventions: Drug: Efavirenz
- INV (Experimental): Indinavir/ritonavir
  Interventions: Drug: Indinavir/ritonavir
- NFV (Experimental): Nelfinavir
  Interventions: Drug: Nelfinavir
- SQV (Experimental): Saquinavir/ritonavir
  Interventions: Drug: Saquinavir/ritonavir
- LPV (Experimental): Lopinavir/ritonavir
  Interventions: Drug: Lopinavir/ritonavir
- ATV (Experimental): Atazanavir
  Interventions: Drug: Atazanavir
- ATV/rtv (Experimental): Atazanavir/ritonavir
  Interventions: Drug: Atazanavir/ritonavir
- Fos-APV (Experimental): Fos-amprenavir/ritonavir
  Interventions: Drug: Fos-amprenavir/ritonavir
- TPV (Experimental): Tipranavir/ritonavir
  Interventions: Drug: Tipranavir/ ritonavir
- DRV (Experimental): Darunavir/ritonavir
  Interventions: Drug: Darunavir/ritonavir

INTERVENTIONS:
Drug: Nevirapine — tablets 200 mg, 400 mg/day
  Other Names: Viramune
  Arms: NVP
Drug: Efavirenz — tablets 600 mg, 600 mg/day
  Other Names: Sustiva
  Arms: EFV
Drug: Indinavir/ritonavir — Indinavir: capsules 400 mg, 1600 mg/day
  Ritonavir: capsules 100 mg, 200 mg/day
  Other Names: Crixivan/norvir
  Arms: INV
Drug: Nelfinavir — tablets 250 mg, 2500 mg/day
  Other Names: Viracept
  Arms: NFV
Drug: Saquinavir/ritonavir — Saquinavir: tablets 500 mg, 2000 mg/day
  Ritonavir: tablets 100 mg, 200 mg/day
  Other Names: Invirase/Norvir
  Arms: SQV
Drug: Lopinavir/ritonavir — tablets lopinavir 200 mg + ritonavir 50 mg, 800/200 mg/day
  Other Names: Kaletra
  Arms: LPV
Drug: Atazanavir — capsules 200 mg, 400 mg/day
  Other Names: Reyataz
  Arms: ATV
Drug: Atazanavir/ritonavir — Atazanavir: capsules 150 mg, 300 mg/day
  Ritonavir: capsules 100 mg, 200 mg/day
  Other Names: Reyataz/Norvir
  Arms: ATV/rtv
Drug: Fos-amprenavir/ritonavir — Fos-amprenavir: capsules 700 mg, 1400 mg/day
  Ritonavir: capsules 100 mg, 200 mg/day
  Other Names: Telzir/norvir
  Arms: Fos-APV
Drug: Tipranavir/ ritonavir — Tipranavir: tablets 250 mg, 1000 mg/day
  Ritonavir: capsules 100 mg, 400 mg/day
  Other Names: Aptivus/Norvir
  Arms: TPV
Drug: Darunavir/ritonavir — Darunavir: tablets 300 mg, 1200 mg/day
  Ritonavir: capsules 100 mg, 200 mg/day
  Other Names: Prezista/norvir
  Arms: DRV

SUMMARY:
The purpose of this study is to characterise the pharmacokinetic profiles of non-nucleoside analog reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs), and the influence of the individual characteristics on the pharmacokinetic parameters in the Spanish population of HIV-infected subjects.

DETAILED DESCRIPTION:
The antiretrovirals were administered conventionally according to fixed dosage systems, or depending on the weight of the individual in the case of certain agents. However, the plasma levels of antiretrovirals following the administration of a fixed dose present a marked interindividual variability. Moreover, a significant proportion of the patients on treatment with PIs presented plasma levels regarded as suboptimal in previous studies.

Moreover, for the correct modification of the dosage of a drug, populational data on its pharmacokinetic behaviour during the dosing interval is required. Only by integrating this information with the specific characteristics of each individual is it possible, using mathematical models, to estimate the effect that a modification of the dosage of the drug would have on its plasma concentration. However, populational data on the pharmacokinetic behaviour of antiretroviral agents are still very limited at this moment, and have not always been obtained in populations similar to the one to which they are to be applied.

Thus, knowing the pharmacokinetic behaviour of the antiretroviral agents in our population and the influence of certain individual characteristics on this behaviour may be of great interest, since only in this way will we be able to tailor the dosage of antiretrovirals reliably in our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age higher than 18 years.
2. Documented HIV infection (at least one positive Western-blot)
3. Stable antiretroviral treatment with PI or NNRTI, no changes over the last 4 weeks.
4. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or negative pregnancy test.

Exclusion Criteria:

1. Subjects on treatment with more than one PI or with combinations of PI and NNRTI (the use of ritonavir in doses below 400 mg BID will not be regarded as a second PI).
2. Treatment with other drugs with known significant pharmacological interactions with the investigational drug over the previous two weeks.
3. Unsuitable adherence to treatment (one or more doses omitted in the last week, or two or more doses omitted in the last two weeks).
4. Presence of clinical findings or a background of gastrointestinal disease or digestive surgery that may interfere in the pharmacokinetics of the medication.
5. Active consumption of alcohol (>50 grams/day) or illegal drugs (except cannabis).
6. In the case of women, pregnancy or breastfeeding.
7. Record or suspicion of inability to cooperate properly

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the plasma concentration of the PI/NNRTI drugs (Ka absorption constant, CI: plasma clearance, Vd: volume of distribution). | In the 12 hour (h) pharmacokinetic curve

SECONDARY OUTCOMES:
Demographic: race, gender, age | In the 12 h pharmacokinetic curve
Clinical: weight, height, liver/renal impairment, HIV infection stage, tobacco/alcohol consumption | In the 12 h pharmacokinetic curve
Adverse events | In the 12 h pharmacokinetic curve
Laboratory: creatinine, albumin, Quick Index, bilirubin, GOT, GPT, GGT, FA, CD4 lymphocyte count, HIV viral load, HBsAg and anti-HCV, alpha acid glycoprotein | In the 12 h pharmacokinetic curve
Antiretroviral and concomitant treatment, adherence (number of doses omitted in the last two weeks) | In the 12 h pharmacokinetic curve
Pharmacokinetics: maximum concentration (Cmax), time to maximum concentration (Tmax), plasma concentration at the end of the posology interval (Ctrough), half-life (T1/2), area under the curve (ABC) | In the 12 h pharmacokinetic curve
Genetic study of polymorphism of CYP3A4 and P-glycoprotein | In the 12 h pharmacokinetic curve

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — Lluita contra la Sida Foundation-HIV Unit
Locations (6):
- Spain (6):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital de Figueres, Figueras, Barcelona
  - Fundació Hospital-Asil de Granollers, Granollers, Barcelona
  - Hospital de Vic, Vic, Barcelona
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

REFERENCES:
- [Derived] Molto J, Xinarianos G, Miranda C, Pushpakom S, Cedeno S, Clotet B, Owen A, Valle M. Simultaneous pharmacogenetics-based population pharmacokinetic analysis of darunavir and ritonavir in HIV-infected patients. Clin Pharmacokinet. 2013 Jul;52(7):543-53. doi: 10.1007/s40262-013-0057-6. PMID 23494984